CLINICAL TRIAL: NCT05180513
Title: Comparing Two Ways to Mitigate the Impact of the COVID-19 Pandemic on Mental Health Among Adults From Underserved and Racial Minority Communities
Brief Title: Mellowing Mind: Comparing Two Technology Based Mindfulness Interventions for Stress Impacted by COVID-19 in Underserved Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Yu-Ping Chang, Principal Investigator, Professor and Associate Dean for Research and Scholarship, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVID-2020C2-1115
Record Dates: First submitted 2021-05-19; First posted 2022-01-06 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Worry; Stress
Keywords: Mindfulness Based Stress Reduction; Community Based Research

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teleconference Mindfulness Intervention Group (Other): MBSR training program that has been adapted for use via Zoom teleconferencing and for cultural relevancy
  Interventions: Behavioral: Teleconference Mindfulness Intervention
- Smartphone App Mindfulness Intervention Group (Other): MBSR training program that has been adapted for use via smartphone app and for cultural relevancy
  Interventions: Behavioral: Smartphone App Mindfulness Intervention
- Waitlist Control Group (No Intervention): No intervention; control group

INTERVENTIONS:
Behavioral: Teleconference Mindfulness Intervention — The teleconference intervention is administered by a trained interventionist via Zoom and is based on a manual adapted from a traditional MBSR version. Practices and activities include meditations, mindful breathing exercises and movements, discussions, and reflections, which participants learn at weekly sessions and practice on their own throughout the week. To adapt the traditional MBSR program for the target community population, intervention materials were reviewed for feedback from community stakeholders, and modified according to their feedback.
  Arms: Teleconference Mindfulness Intervention Group
Behavioral: Smartphone App Mindfulness Intervention — The smartphone app intervention is administered through the app. The smartphone app aligns with the traditional MBSR format, but training and practice is done individually and independently by members of this group. To adapt the traditional MBSR program for the target community population, the app was tested by community stakeholders and modified according to their feedback.
  Arms: Smartphone App Mindfulness Intervention Group

SUMMARY:
The purpose of this study is to examine the comparative effectiveness of two technology-based Mindfulness Based Stress Reduction (MBSR) programs (one via video/teleconference and one via a smartphone app) for reducing worry, anxiety and/or related mental health effects of stress in members of identified underserved communities, which were highly impacted by the COVID-19 pandemic.

DETAILED DESCRIPTION:
The purpose of this randomized controlled study is to examine the comparative effectiveness of two technology-based Mindfulness Based Stress Reduction (MBSR) programs (one via video/teleconference and one via a smartphone app) for reducing worry, anxiety, and/or related mental health effects of stress in members of identified underserved communities, which were highly impacted by the COVID-19 pandemic. Participants will be randomly assigned to a teleconference MBSR program, a MBSR smartphone app program, or a waitlist control group. Each intervention includes participation in a 9-week (8 sessions plus an introduction) mindfulness intervention that consists of instruction and daily practice. Questionnaires and semi-structured interviews will be administered at mid-intervention, post-intervention, and one-month and three-month follow-up points. It is hypothesized that participants in the two intervention groups will show measurable and sustained improvement in the primary outcome, worry, as well as in the secondary outcomes, anxiety and related mental health effects. It is further hypothesized that the smartphone app mindfulness intervention will show similar effectiveness to the teleconference mindfulness intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Significant worry as per the Penn State Worry Questionnaire-Abbreviated [PSWQ-A]
* Fluent in English
* Reside in one of the local city zip codes, identified as underserved, and primarily African American, communities

Exclusion Criteria:

* Severe depression as per Patient Health Questionnaire [PHQ-9]
* Active suicidal intent as per PHQ-9 question 9
* Diagnosis of psychosis, or bipolar disorder, or moderate or severe substance use disorder in the past month as per self report
* Cognitive impairment as per (modified) Short Portable Mental Status Questionnaire [SPMSQ]
* Currently receiving psychotherapy or behavioral counseling, including MBSR
* Change in psychotropic medications within the last month as per self report
* Unable to communicate in a way that would allow for participation in screenings or sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Worry from baseline to mid-intervention at five weeks, post-intervention at nine weeks, and follow-ups to assess sustainability at one and three months following end of intervention | 21 Weeks: Change from Baseline score to score at mid-intervention, post-intervention, and follow-up scores at one month and three months past end of intervention
  A total score on the Penn State Worry Questionnaire [PSWQ], a scaled measure with total scores ranging from 16 to 80, in which higher scores indicate greater severity of worry

SECONDARY OUTCOMES:
Changes in Anxiety from baseline to mid-intervention at five weeks, post-intervention at nine weeks, and follow-ups to assess sustainability at one and three months following end of intervention | 21 Weeks: Change from Baseline score to score at mid-intervention, post-intervention, and follow-up scores at one month and three months past end of intervention
  A total score on the Generalized Anxiety Disorder Scale [GAD-7], a scaled measure with total scores ranging from 0 to 21, in which higher scores indicate more severe anxiety
Changes in Perceived Stress from baseline to mid-intervention at five weeks, post-intervention at nine weeks, and follow-ups to assess sustainability at one and three months following end of intervention | 21 Weeks: Change from Baseline score to score at mid-intervention, post-intervention, and follow-up scores at one month and three months past end of intervention
  A total score on the Perceived Stress Scale [PSS], a scaled measure with total scores ranging from 0 to 40, in which higher scores indicate higher levels of perceived stress
Changes in Depression from baseline to mid-intervention at five weeks, post-intervention at nine weeks, and follow-ups to assess sustainability at one and three months following end of intervention | Change from Baseline score to score at mid-intervention, post-intervention, and follow-up scores at one month and three months past end of intervention
  A total score on the Patient Health Questionnaire [PHQ-9], a scaled measure for assessing minimal to severe depression, with total scores ranging from 0 to 27, in which higher scores indicate more severe depression
Changes in Sleep Quality from baseline to mid-intervention at five weeks, post-intervention at nine weeks, and follow-ups to assess sustainability at one and three months following end of intervention | 21 weeks Change from Baseline score to score at mid-intervention, post-intervention, and follow-up scores at one month and three months past end of intervention
  A global score on the Pittsburgh Sleep Quality Index [PSQI], which contains seven scaled components for sleep quality, with global scores ranging from 0 to 21, in which lower global scores indicate better overall quality of sleep.
Changes in Loneliness from baseline to mid-intervention at five weeks, post-intervention at nine weeks, and follow-ups to assess sustainability at one and three months following end of intervention | 21 Weeks Change from Baseline score to score at mid-intervention, post-intervention, and follow-up scores at one month and three months past end of intervention
  A total score on the UCLA Loneliness Scale, a scaled measure with total scores ranging from 0 to 60, in which higher total scores indicate higher levels of loneliness
Changes in Social Disconnectedness from baseline to mid-intervention at five weeks, post-intervention at nine weeks, and follow-ups to assess sustainability at one and three months following end of intervention | 21 Weeks Change from Baseline score to score at mid-intervention, post-intervention, and follow-up scores at one month and three months past end of intervention
  A total score on the Social Disconnectedness Scale, a scaled measure with total scores ranging from 0 to 43, in which higher scores indicate higher social disconnectedness
Changes in Mindfulness from baseline to mid-intervention at five weeks, post-intervention at nine weeks, and follow-ups to assess sustainability at one and three months following end of intervention | 21 weeks Change from Baseline score to score at mid-intervention, post-intervention, and follow-up scores at one month and three months past end of intervention
  A global score on the Five Facet Mindfulness Questionnaire [FFMQ], which contains five scaled components for attributes of mindfulness and with total scores ranging from 39 to 195, in which higher global scores indicate greater overall mindfulness
Quality of life, satisfaction with | 21 Weeks Change from Baseline score to score at mid-intervention, end of intervention, and follow-up scores at one month and three months past end of intervention
  A total score on the Quality of Life Scale [QOLS], a scaled measure with total scores ranging from16 to 112, in which higher total scores indicate greater satisfaction with or quality of life
Changes in Psychological Well-being from baseline to mid-intervention at five weeks, post-intervention at nine weeks, and follow-ups to assess sustainability at one and three months following end of intervention | 21 Weeks Change from Baseline score to score at mid-intervention, post-intervention, and follow-up scores at one month and three months past end of intervention
  A total score on the Flourishing Scale [FS], a scaled measure with with total scores ranging from 8 to 56, in which higher total scores indicate greater flourishing or psychological well-being

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ping Chang, PhD, Principal Investigator — SUNY at Buffalo School of Nursing
Locations (1):
- State University of New York, University at Buffalo, Buffalo, New York, United States